CLINICAL TRIAL: NCT02975934
Title: TRITON3: A Multicenter, Randomized, Open Label Phase 3 Study of Rucaparib Versus Physician's Choice of Therapy for Patients With Metastatic Castration Resistant Prostate Cancer Associated With Homologous Recombination Deficiency
Brief Title: A Study of Rucaparib Versus Physician's Choice of Therapy in Participants With Metastatic Castration-resistant Prostate Cancer and Homologous Recombination Gene Deficiency
Acronym: TRITON3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-063; 2016-003163-20 (EudraCT Number)
Record Dates: First submitted 2016-11-19; First posted 2016-11-29 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: CRPC; PARP inhibitor; PARPi; BRCA; ATM; HRD; TRITON; homologous recombination; DNA repair; DNA defect; DNA anomaly; germline; somatic; mCRPC
MeSH Terms: interventions — rucaparib; Abiraterone Acetate; enzalutamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rucaparib (Experimental): Oral rucaparib (monotherapy).
  Interventions: Drug: Rucaparib
- Abiraterone acetate or Enzalutamide or Docetaxel (Active Comparator): Oral abiraterone acetate (monotherapy, given in combination with prednisone). Oral enzalutamide (monotherapy). Intravenous docetaxel (monotherapy, given in combination with prednisone or prednisolone).
  Interventions: Drug: Abiraterone acetate or Enzalutamide or Docetaxel

INTERVENTIONS:
Drug: Rucaparib — Rucaparib will be administered daily.
  Other Names: CO-338
  Arms: Rucaparib
Drug: Abiraterone acetate or Enzalutamide or Docetaxel — Abiraterone acetate and enzalutamide will be administered daily. Docetaxel will be administered every 3 weeks.
  Other Names: Zytiga (abiraterone acetate) or Xtandi (enzalutamide) or Taxotere (docetaxel)
  Arms: Abiraterone acetate or Enzalutamide or Docetaxel

SUMMARY:
The purpose of this study is to determine how participants with metastatic castration-resistant prostate cancer, and evidence of a homologous recombination gene deficiency, respond to treatment with rucaparib versus treatment with physician's choice of abiraterone acetate, enzalutamide, or docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old at the time the informed consent is signed
* Have a histologically or cytologically confirmed adenocarcinoma or poorly differentiated carcinoma of the prostate that is metastatic
* Be surgically or medically castrated, with serum testosterone levels of ≤ 50 ng/dL (1.73 nM)
* Be eligible for treatment with physician's choice of comparator treatment (abiraterone acetate, enzalutamide or docetaxel)
* Experienced disease progression after having received 1 prior next generation androgen receptor-targeted therapy
* Have a deleterious mutation in a BRCA1/2 or ATM gene

Exclusion Criteria:

* Active second malignancy, with the exception of curatively treated non melanoma skin cancer, carcinoma in situ, or superficial bladder cancer
* Prior treatment with any PARP inhibitor
* Prior treatment with chemotherapy for metastatic castration-resistant prostate cancer
* Symptomatic and/or untreated central nervous system metastases
* Pre-existing duodenal stent and/or any gastrointestinal disorder or defect that would, in the opinion of the investigator, interfere with absorption of study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (150):
- United States (61):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Arizona Oncology Associates - USOR, Tucson, Arizona
  - University of Southern California, Beverly Hills, California
  - Alliance Research Centers, Laguna Hills, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - San Bernardino Urological Associates, San Bernardino, California
  - Sharp Memorial Hospital, San Diego, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - San Francisco VA Health Care System, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Kaiser Permanente, Northern CA, Vallejo, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Medical Oncology Hematology Consultants - USOR, Newark, Delaware
  - Boca Raton Community Hospital, Inc., Boca Raton, Florida
  - University of Florida Health Cancer Center, Orlando, Florida
  - Atlanta Urological Group, Atlanta, Georgia
  - Kaiser Permanente Medical Group, Honolulu, Hawaii
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Maryland Oncology Hematology P.A., Columbia, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Minnesota Veterans Research Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, MN, Rochester, Minnesota
  - Alegent Health Bergan Mercy Hospital , GU Research Network, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Premier Urology Associates, Lawrenceville, New Jersey
  - Roswell Park, Buffalo, New York
  - NYU Perlmutter Cancer Center, New York, New York
  - Memorial Sloan Kettering CC, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina Lineberger Cancer Center, Chapel Hill, North Carolina
  - Carolina Urology Partners, Concord, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - The Urology Group, Cincinnati, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - VA Portland Health Care System, Portland, Oregon
  - Northwest Cancer Specialist DBA Compass Oncology, Portland, Oregon
  - Knight Cancer Institute, Portland, Oregon
  - Urology Associates Clinical Research, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Health Science Center, Houston, Texas
  - Texas Oncology Cancer Center-Round Rock, Round Rock, Texas
  - Urology of Virginia, Virginia Beach, Virginia
  - MultiCare Regional Cancer Center - Gig Harbor, Gig Harbor, Washington
  - VA Puget Sound HCS, Seattle, Washington
  - University of Washington Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (8):
  - Southside Cancer Care Centre, Miranda, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Northern Cancer Insitute, St. Leonards, Saint Leonards, New South Wales
  - St John of God Hospital, Subiaco, Subiaco, Western Australia
  - Peninsula & Southeast Oncology, Frankston
  - Barwon Health, University Hospital Geelong, Geelong
  - Royal Hobart Hospital, Hobart
  - Riverina Cancer Care Centre, Wagga Wagga
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - AZ Groeninge, Kortrijk
  - CHU Sart-Tilman, Liège
  - Clinique et Maternité Sainte-Elisabeth, Namur
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Centre Hospitalier Universitaire Dr-Georges-L.-Dumont, Moncton, New Brunswick
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Lakeridge Health Medical Specialty Medical Oncology, Oshawa
  - Sunnybrook Odette Cancer Centre, Toronto
- Denmark (3):
  - Copenhagen University Hospital, Copenhagen
  - Herlev Hospital, Herlev
  - Vejle Sygehus, Vejle
- France (9):
  - Centre Georges François Leclerc, Dijon
  - Clinique Victor Hugo Centre Jean Bernard, Le Mans
  - Hôpital Privé La Louvière, Lille
  - Centre Léon Bérard, Lyon
  - Polyclinique de Gentilly (Centre D'Oncologie De Gentilly), Nancy
  - Institut Curie, Paris
  - Centre Armoricain de Radiotherapie, Imagerie medicale et Oncologie, CARIO, Plérin
  - CRLCC Eugene Marquis, Rennes
  - Institut Gustave-Roussy, Villejuif
- Germany (14):
  - Gemeinschaftspraxis für Hämatologie&Onkologie, Augsburg
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Apotheke des Städtischen Klinikums Braunschweig, Braunschweig
  - Universitätsklinikum Köln, Cologne
  - University Hospital Carl Gustav Carus, Dresden
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Urologische Gemeinschaftspraxis, Emmendingen
  - Universitaetsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Universitatsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Medizinischen Fakultät Mannheim der Universität Heidelberg, Mannheim
  - Studienpraxis Urologie, Nürtingen
  - University of Tuebingen, Tübingen
  - Die GesundheitsUnion (DGU), Wuppertal
- Ireland (6):
  - Cork University Hospital, Cork
  - Adelaide & Meath Hospital, Incorporating the National Children's Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital (MPH), Dublin
  - St James's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
- Israel (6):
  - Rambam Health Care Campus (RHCC), Rambam Medical Center, Haifa
  - Hadassah University Hospital, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - The Tel Aviv Sourasky Medical Center (Ichilov Hospital), Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (8):
  - Ospedale San Donato, Azienda USLSUDEST, Arezzo
  - Ospedale Santa Maria delle Croci, Faenza
  - Romagnolo per lo Studio e la Cura dei Tumori IRST-IRCCS - Oncologia medica, Meldola
  - IEO Instituto Europeo di Oncologia, Milan
  - University of Modena and Reggio Emilia, Modena
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Azienda Opsedaliera S. Maria di Terni, Terni
  - Presidio Ospedaliero Santa Chiara di Trento, Trento
- Spain (14):
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Hospital Universitario Lucus Augusti., Lugo
  - MD Anderson Cancer Center - Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Marques de Valdecilla University Hospital (HUMV), Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Instituto Valenciano de Oncología, Valencia
- United Kingdom (9):
  - Guy's and St Thomas' NHS Foundation Trust, London, England
  - Royal Marsden Hospital, London, England
  - Oxford Cancer Centre, Medical Oncology Unit, Oxford, England
  - Royal Preston Hospital, Preston, England
  - Wexham Park Hospital, Slough, England
  - Velindre Hospital, Cardiff
  - Royal Marsden Hospital, London
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets for study results will be made available to qualified researchers in compliance with applicable privacy laws and data protection regulations.
  Data will be provided by pharmaand GmbH.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available to qualified researchers after the primary, secondary, and/or exploratory outcomes of the study are reported or published and for 1 year thereafter.
Access Criteria: Requests for de-identified datasets will be made available to qualified researchers following submission of a methodologically sound proposal to medinfo@pharmaand.com.

REFERENCES:
- [Result] Fizazi K, Piulats JM, Reaume MN, Ostler P, McDermott R, Gingerich JR, Pintus E, Sridhar SS, Bambury RM, Emmenegger U, Lindberg H, Morris D, Nole F, Staffurth J, Redfern C, Saez MI, Abida W, Daugaard G, Heidenreich A, Krieger L, Sautois B, Loehr A, Despain D, Heyes CA, Watkins SP, Chowdhury S, Ryan CJ, Bryce AH; TRITON3 Investigators. Rucaparib or Physician's Choice in Metastatic Prostate Cancer. N Engl J Med. 2023 Feb 23;388(8):719-732. doi: 10.1056/NEJMoa2214676. Epub 2023 Feb 16. PMID 36795891
- [Derived] Collins K, Cheng L. Reprint of: morphologic spectrum of treatment-related changes in prostate tissue and prostate cancer: an updated review. Hum Pathol. 2023 Mar;133:92-101. doi: 10.1016/j.humpath.2023.02.007. Epub 2023 Mar 8. PMID 36898948
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate or Enzalutamide or Docetaxel: Oral abiraterone acetate (monotherapy, given in combination with prednisone). Oral enzalutamide (monotherapy). Intravenous docetaxel (monotherapy, given in combination with prednisone or prednisolone).
  Abiraterone acetate or Enzalutamide or Docetaxel: Abiraterone acetate and enzalutamide will be administered daily.
  Docetaxel will be administered every 3 weeks.
- Rucaparib (Cross-Over Phase): Oral rucaparib (monotherapy).
  Rucaparib: Rucaparib will be administered daily. Participants from the Abiraterone Acetate/Enzalutamide/Docetaxel arm who completed the Treatment Phase and radiographically progressed by independent radiology review (IRR) may receive rucaparib treatment during the Cross-Over Phase.
  After analysis of the primary endpoint, investigator-assessed radiographic disease progression will be used for cross-over eligibility evaluation.
Period: Treatment Phase
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel | Rucaparib (Cross-Over Phase)
Started | 270 | 135 | 0
Received at Least 1 Dose of Study Drug | 270 | 130 | 0
Safety Population | 270 | 130 | 0
Completed (Treatment period completion was defined as discontinuation when criteria for treatment discontinuation were met.) | 270 | 130 | 0
Not Completed | 0 | 5 | 0
Not completed — Never initiated study drug | 0 | 5 | 0
Period: Cross-Over Phase
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel | Rucaparib (Cross-Over Phase)
Started | 0 | 0 | 70
Received at Least 1 Dose of Study Drug | 0 | 0 | 70
Safety Population | 0 | 0 | 70
Completed (Crossover period completion was defined as discontinuation when criteria for treatment discontinuation were met, or study closure.) | 0 | 0 | 70
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all randomized participants (participants with breast cancer gene [BRCA] mutated metastatic castration-resistant prostate cancer [mCRPC] and participants with ataxia- telangiectasia mutated serine/threonine kinase [ATM] mutated mCRPC).
Groups:
- Total: Total of all reporting groups
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel | Total
Number analyzed (Participants) | 270 | 135 | 405
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 32 | 116
  >=65 years | 186 | 103 | 289
Age, Continuous [Median (Full Range); unit: years] | 70 [45 to 90] | 71 [47 to 92] | 70 [45 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 270 | 135 | 405
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 216 | 103 | 319
  Unknown or Not Reported | 51 | 28 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 4 | 14
  White | 199 | 103 | 302
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 53 | 27 | 80
Region of Enrollment [Number; unit: participants]
  North America | 111 | 56 | 167
  Europe | 141 | 73 | 214
  Australia | 10 | 3 | 13
  Israel | 8 | 3 | 11
ECOG Performance Status (at stratification) [Count of Participants; unit: Participants] — Measure Description: Eastern Cooperative Oncology Group (ECOG) Performance Status Scale. ECOG 0 = Fully active, able to carry on all pre-disease performance without restriction. ECOG 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (eg, light house work or office work)
  Participants
    0 | 132 | 68 | 200
    1 | 138 | 67 | 205
Gene Alteration (at stratification) [Count of Participants; unit: Participants]
  BRCA1 | 29 | 15 | 44
  BRCA2 | 172 | 86 | 258
  ATM | 69 | 34 | 103
Baseline prostate specific antigen (PSA) [Median (Full Range); unit: ng/ml] | 26.9 [0.1 to 1247] | 28.8 [0 to 1039] | 27.8 [0 to 1247]
Gleason score ≥8 at diagnosis [Count of Participants; unit: Participants] — The scale for the Gleason score ranges from 2 to 10, with higher scores indicating a worse prognosis
  Participants | 173 | 96 | 269
Measurable Disease per Independent Radiological Review (IRR) [Count of Participants; unit: Participants] | 106 | 55 | 161
Metastases site(s) by IRR [Count of Participants; unit: Participants] — Participants may be counted in more than one category
  Participants
    Bone | 235 | 114 | 349
    Nodal | 118 | 60 | 178
    Visceral | 74 | 46 | 120
Prior Therapies for CRPC [Count of Participants; unit: Participants]
  0 | 48 | 26 | 74
  ≥1 | 222 | 109 | 331
Prior therapy (2nd generation androgen receptor pathway inhibitor (ARPI) or docetaxel only) [Count of Participants; unit: Participants] — Participants may be counted in more than one category
  Participants
    Abiraterone acetate | 150 | 80 | 230
    Apalutamide | 8 | 1 | 9
    Enzalutamide | 119 | 61 | 180
    Docetaxel for hormone-sensitive prostate cancer | 63 | 28 | 91

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-free Survival (rPFS) by IRR in Participants With a BRCA Alteration
Description: The primary efficacy endpoint for the study is rPFSirr, defined as the time from randomization to the first objective evidence of radiographic progression, or death due to any cause (whichever occurs first).
  Radiographic disease progression includes confirmed soft tissue disease progression and confirmed bone disease progression as per modified RECIST Version 1.1 (at least a 20% increase in the sum of the LD of target lesions or appearance of one or more new extra-skeletal lesions and/or unequivocal progression of existing nontarget lesions) or PCWG3 criteria Progression by bone is determined by PCWG3 criteria in which at least two new lesions appearing during the first 12-week flare window followed by 2 additional new lesions in the confirmatory scan appearing after the 12-week flare window, or after the 12-week flare window, at least 2 new lesions relative to the first post-treatment scan confirmed on a subsequent scan).
Time Frame: From enrollment to primary completion of study (Total follow-up was up to approximately 4 years)
Population: ITT Population with BRCA mutated mCRPC.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 201 | 101
months | 11.2 [9.2 to 13.8] | 6.4 [5.4 to 8.3]
Statistical Analysis 1: Comparison: Rucaparib vs Abiraterone Acetate or Enzalutamide or Docetaxel; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.36 to 0.69]

2. Primary Outcome: Radiographic Progression-free Survival (rPFS) by IRR in Participants With a BRCA or ATM Alteration Combined
Description: The primary efficacy endpoint for the study is rPFSirr, defined as the time from randomization to the first objective evidence of radiographic progression, or death due to any cause (whichever occurs first).
  Radiographic disease progression includes confirmed soft tissue disease progression and confirmed bone disease progression as per modified RECIST Version 1.1 (at least a 20% increase in the sum of the LD of target lesions or appearance of one or more new extra-skeletal lesions and/or unequivocal progression of existing nontarget lesions) or PCWG3 criteria (Progression by bone is determined by PCWG3 criteria in which at least two new lesions appearing during the first 12-week flare window followed by 2 additional new lesions in the confirmatory scan appearing after the 12-week flare window, or after the 12-week flare window, at least 2 new lesions relative to the first post-treatment scan confirmed on a subsequent scan).
Time Frame: From enrollment to primary completion of study (Total follow-up was up to approximately 4 years)
Population: ITT Population included all randomized participants (participants with BRCA mutated mCRPC and participants with ATM mutated mCRPC).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 270 | 135
months | 10.2 [8.3 to 11.2] | 6.4 [5.6 to 8.2]
Statistical Analysis 1: Comparison: Rucaparib vs Abiraterone Acetate or Enzalutamide or Docetaxel; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.47 to 0.80]

3. Secondary Outcome: Overall Survival in Participants With a BRCA Alteration
Description: Overall survival time is calculated as the time from randomization to death (by any cause) +1 day. Participants who have not died will be censored on the date the participant was last known to be alive.
Time Frame: From enrollment to completion of study (up to approximately 7 years)
Population: ITT Population with BRCA mutated mCRPC.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 201 | 101
months | 23.2 [19.1 to 25.2] | 21.2 [18.0 to 23.1]
Statistical Analysis 1: Comparison: Rucaparib vs Abiraterone Acetate or Enzalutamide or Docetaxel; Test type: Superiority; p = 0.5044, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.68 to 1.20]

4. Secondary Outcome: Overall Survival in Participants With a BRCA or ATM Alteration Combined
Description: Overall survival time is calculated as the time from randomization to death (by any cause) +1 day. Participants who have not died will be censored on the date the participants was last known to be alive.
Time Frame: From enrollment to completion of study (up to approximately 7 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 270 | 135
months | 22.8 [19.0 to 24.2] | 21.7 [18.9 to 23.3]
Statistical Analysis 1: Comparison: Rucaparib vs Abiraterone Acetate or Enzalutamide or Docetaxel; Test type: Superiority; p = 0.9368, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.78 to 1.26]

5. Secondary Outcome: Objective Response Rate (ORR) by IRR in Participants With a BRCA Alteration
Description: ORR is defined as the percentage of participants with a confirmed best response of Complete response (CR) or Partial Response (PR) in participants with measurable disease at study entry. Modified RECIST Version 1.1 criteria is used to determine ORR (ie, CR or PR by IRR assessment and no progression in bone per PCWG3 by IRR assessment).
  CR is disappearance of all target and non-target lesions; any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From enrollment to primary completion of study (Total follow-up was up to approximately 4 years)
Population: ITT Population with BRCA mutated mCRPC and measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 82 | 41
Participants | 37 | 7

6. Secondary Outcome: Objective Response Rate (ORR) by IRR in Participants With a BRCA or ATM Alteration Combined
Description: as for outcome 5
Time Frame: From enrollment to primary completion of study (Total follow-up was up to approximately 4 years)
Population: ITT Population included all randomized participants (participants with BRCA mutated mCRPC and participants with ATM mutated mCRPC) with measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 106 | 55
Participants | 37 | 9

7. Secondary Outcome: Duration of Response (DOR) by IRR in Participants With a BRCA Alteration
Description: DOR is defined as the time from the first confirmed response (CR or PR by modified RECIST Version 1.1 in participants with nodal or visceral ± nodal disease) until the first date that Progressive Disease (PD) (using the same criteria) is documented.
Time Frame: From enrollment to primary completion of study (Total follow-up was up to approximately 4 years)
Population: ITT Population with BRCA mutated mCRPC and measurable disease at baseline. 'Overall number of participants analyzed' = participants with objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 37 | 7
months | 7.4 [6.4 to 12.7] | 7.4 [3.5 to NA] — The upper limit of the confidence interval is inestimable likely due to the small number of participants in this treatment group.

8. Secondary Outcome: Duration of Response (DOR) by IRR in Participants With a BRCA or ATM Alteration Combined
Description: as for outcome 7
Time Frame: From enrollment to primary completion of study (Total follow-up was up to approximately 4 years)
Population: ITT Population included all randomized participants (participants with BRCA mutated mCRPC and participants with ATM mutated mCRPC) with measurable disease at baseline. 'Overall number of participants analyzed' = participants with objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 37 | 9
months | 7.4 [6.4 to 12.7] | 7.4 [3.5 to 14.5]

9. Secondary Outcome: PSA Response in Participants With a BRCA Alteration
Description: Confirmed PSA response is defined as ≥ 50% reduction in PSA from baseline on at least two assessments conducted at least 3 weeks apart. PSA response is calculated for all participants with PSA values at baseline and at least one post-baseline assessment. PSA is assessed by a local laboratory.
Time Frame: From enrollment to primary completion of study (up to approximately 5 years)
Population: ITT Population with BRCA mutated mCRPC.
Measure: Number; unit: percentage of participants
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 201 | 101
percentage of participants | 54.7 | 26.7

10. Secondary Outcome: PSA Response in Participants With a BRCA or ATM Alteration Combined
Description: as for outcome 9
Time Frame: From enrollment to primary completion of study (up to approximately 5 years)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 270 | 135
percentage of participants | 41.9 | 26.7

11. Secondary Outcome: Clinical Benefit Rate (CBR) by IRR at 6 Months in Participants With a BRCA Alteration
Description: Defined as the percentage of participants with a complete response (CR), partial response (PR), and stable disease (SD) according to modified RECIST Version 1.1 with no progression in bone per PCWG3 criteria.
Time Frame: From enrollment to 6 months
Population: The Safety Population included all participants with BRCA mutated mCRPC who received at least one dose of protocol-specified treatment and had 6 months of follow-up prior to the data cutoff.
Measure: Number; unit: percentage of participants
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 200 | 97
percentage of participants | 63.0 | 22.7

12. Secondary Outcome: Clinical Benefit Rate (CBR) by IRR at 6 Months in Participants With a BRCA or ATM Alteration Combined
Description: Defined as the percentage of participants with a Complete Response (CR), Partial Response (PR), and Stable Disease (SD), according to Modified RECIST Version 1.1 with no progression in bone per PCWG3 Criteria.
Time Frame: From enrollment to 6 months
Population: The Safety Population included all participants who received at least one dose of protocol-specified treatment and had 6 months of follow-up prior to the data cutoff.
Measure: Number; unit: percentage of participants
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 269 | 130
percentage of participants | 57.6 | 25.4

13. Secondary Outcome: Time to Prostate Specific Antigen (PSA) Progression in Participants With a BRCA Alteration
Description: Time to PSA progression is defined as the time from randomization to the date that a ≥ 25% increase and absolute increase of ≥ 2 ng/mL above the nadir (or baseline value for participants who did not have a decline in PSA) in PSA was measured. The increase must be confirmed by a second consecutive assessment conducted at least 3 weeks later.
Time Frame: From enrollment to primary completion of study (up to approximately 5 years)
Population: ITT Population with BRCA mutated mCRPC.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 201 | 101
months | 6.6 [5.9 to 7.7] | 3.8 [3.1 to 4.5]

14. Secondary Outcome: Time to Prostate Specific Antigen (PSA) Progression in Participants With a BRCA or ATM Alteration Combined
Description: as for outcome 13
Time Frame: From enrollment to primary completion of study (up to approximately 5 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 270 | 135
months | 5.7 [4.6 to 6.5] | 3.6 [3.2 to 4.5]

15. Secondary Outcome: Change in Patient-reported Outcome (PRO) in Participants With a BRCA Alteration: FACT-P
Description: Changes in health and pain status from baseline to week 25 using: Functional Assessment of Cancer Therapy-Prostate questionnaire (FACT-P total score, on a scale of 0 to 156 where a higher score is better quality of life). The greater the decrease in score (ie more negative) from baseline to week 25 the greater the decrease in health status. Assessments completed during screening, at study treatment visits (Day 1, Day 15, Day 29, Day 43, Day 57, and every 29 days thereafter) (during the Treatment Phase, the Treatment Discontinuation Visit, and during the Follow-up Phase.
Time Frame: From enrollment to up to approximately 25 weeks
Population: ITT Population with BRCA mutated mCRPC. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 136 | 35
units on a scale | -0.8 (1.13) | -3.9 (2.23)

16. Secondary Outcome: Change in Patient-reported Outcome (PRO) in Participants With a BRCA Alteration: BPI-SF
Description: Changes in health and pain status from baseline to week 25 using: Brief Pain Inventory-Short Form (BPI-SF) questionnaire (on a scale of 1 to 10, from mild to severe, for pain and pain-interference scores). A decrease indicates less severe pain/interference. Assessments completed during screening, at study treatment visits (Day 1, Day 15, Day 29, Day 43, Day 57, and every 29 days thereafter) (during the Treatment Phase, the Treatment Discontinuation Visit, and during the Follow-up Phase.
Time Frame: From enrollment to up to approximately 25 weeks
Population: ITT Population with BRCA mutated mCRPC. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for specified category.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 133 | 32
units on a scale
  BPI-SF Pain Score | -0.32 (0.139) | 0.14 (0.285)
  BPI-SF Interference Score: number analyzed (Participants) | 130 | 31
  BPI-SF Interference Score | -0.28 (0.147) | 0.65 (0.302)

17. Secondary Outcome: Change in Patient-reported Outcome (PRO) in Participants With a BRCA Alteration: EQ-5D-5L
Description: Changes in health and pain status from baseline to week 25 using: EuroQol-5D-5L Visual Analogue Scale (EQ-5D-5L VAS; on a scale from 100 to 0, from best to worst health status). The greater the increase in score (including more negative) from baseline to week 25 the greater the increase in health status. Assessments completed during screening, at study treatment visits (Day 1, Day 15, Day 29, Day 43, Day 57, and every 29 days thereafter) during the Treatment Phase, the Treatment Discontinuation Visit, and during the Follow-up Phase.
Time Frame: From enrollment to up to approximately 25 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rucaparib | Abiraterone Acetate or Enzalutamide or Docetaxel
Number analyzed (Participants) | 136 | 36
units on a scale | 2.4 (1.23) | 1.8 (2.39)

18. Secondary Outcome: Trough Plasma PK (Cmin) of Rucaparib Based on Sparse Sampling
Description: Mean trough PK plasma concentration over time in the safety population with at least one PK sample collected at timepoints week 5, 9, 13 and 17; only Week 5 data presented.
Time Frame: From enrollment to week 5 of dosing
Population: Safety Population with at least 1 PK sample collected.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Rucaparib
Number analyzed (Participants) | 228
ng/mL | 1310 [5.5 to 4180]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 28 days after receiving the last dose of study drug (approximately 7 years).
Description: All-Cause Mortality is reported for the ITT population. SAEs and AEs were assessed in the Safety Population. After 28 days following last dose of study drug, only SAEs assessed as potentially related to study drug are reported. Events of progression of the participant's underlying cancer, events clearly related to progression of the participant's cancer and progression of disease leading to death are not reported as an AE or SAE.
Groups:
- Rucaparib (Treatment Phase): Oral rucaparib (monotherapy).
  Rucaparib: Rucaparib will be administered daily.
- Abiraterone Acetate or Enzalutamide or Docetaxel (Treatment Phase): Oral abiraterone acetate (monotherapy, given in combination with prednisone). Oral enzalutamide (monotherapy). Intravenous docetaxel (monotherapy, given in combination with prednisone or prednisolone).
  Abiraterone acetate or Enzalutamide or Docetaxel: Abiraterone acetate and enzalutamide will be administered daily.
  Docetaxel will be administered every 3 weeks.
Arm/Group | Rucaparib (Treatment Phase) | Abiraterone Acetate or Enzalutamide or Docetaxel (Treatment Phase) | Rucaparib (Cross-over Phase)
All-Cause Mortality (participants affected / at risk) | 6/270 | 3/135 | 1/70
Serious Adverse Events (participants affected / at risk) | 81/270 | 36/130 | 18/70
Other Adverse Events (participants affected / at risk) | 270/270 | 127/130 | 67/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rucaparib (Treatment Phase) (N=270) | Abiraterone Acetate or Enzalutamide or Docetaxel (Treatment Phase) (N=130) | Rucaparib (Cross-over Phase) (N=70)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 0 (0) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 8 (11) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (2) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blastocystis infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dermo-hypodermitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 1 (2) | 3 (3)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (10) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (3) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sacral radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 8 (9) | 0 (0) | 2 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (3) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rucaparib (Treatment Phase) (N=270) | Abiraterone Acetate or Enzalutamide or Docetaxel (Treatment Phase) (N=130) | Rucaparib (Cross-over Phase) (N=70)
Anaemia (Blood and lymphatic system disorders) | 121 (435) | 24 (30) | 26 (90)
Neutropenia (Blood and lymphatic system disorders) | 17 (37) | 6 (6) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 24 (44) | 0 (0) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 21 (23) | 10 (11) | 3 (6)
Abdominal pain upper (Gastrointestinal disorders) | 15 (15) | 3 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 76 (101) | 19 (23) | 12 (16)
Diarrhoea (Gastrointestinal disorders) | 85 (118) | 36 (49) | 10 (11)
Dyspepsia (Gastrointestinal disorders) | 18 (25) | 5 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 137 (222) | 25 (44) | 26 (41)
Stomatitis (Gastrointestinal disorders) | 12 (20) | 10 (15) | 0 (0)
Vomiting (Gastrointestinal disorders) | 65 (98) | 11 (16) | 12 (25)
Asthenia (General disorders) | 58 (136) | 20 (36) | 9 (12)
Fatigue (General disorders) | 117 (203) | 63 (123) | 23 (41)
Oedema peripheral (General disorders) | 55 (70) | 21 (29) | 14 (15)
Pyrexia (General disorders) | 15 (17) | 7 (11) | 6 (6)
COVID-19 (Infections and infestations) | 16 (17) | 5 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 20 (29) | 3 (3) | 7 (11)
Contusion (Injury, poisoning and procedural complications) | 11 (11) | 7 (7) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 15 (22) | 6 (7) | 3 (3)
Alanine aminotransferase increased (Investigations) | 67 (146) | 3 (3) | 19 (44)
Aspartate aminotransferase increased (Investigations) | 65 (120) | 4 (5) | 20 (46)
Blood alkaline phosphatase increased (Investigations) | 17 (19) | 2 (2) | 2 (3)
Blood bilirubin increased (Investigations) | 13 (43) | 1 (1) | 7 (17)
Blood creatinine increased (Investigations) | 55 (97) | 6 (8) | 8 (10)
Lymphocyte count decreased (Investigations) | 11 (27) | 7 (10) | 4 (9)
Neutrophil count decreased (Investigations) | 17 (64) | 5 (5) | 4 (11)
Platelet count decreased (Investigations) | 29 (103) | 0 (0) | 4 (20)
Weight decreased (Investigations) | 40 (65) | 15 (21) | 10 (18)
White blood cell count decreased (Investigations) | 18 (52) | 3 (7) | 7 (27)
Decreased appetite (Metabolism and nutrition disorders) | 99 (139) | 29 (43) | 18 (27)
Dehydration (Metabolism and nutrition disorders) | 9 (9) | 3 (4) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 17 (51) | 4 (5) | 3 (16)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (16) | 10 (17) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 19 (34) | 7 (13) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 52 (69) | 28 (41) | 9 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 65 (97) | 26 (31) | 13 (19)
Bone pain (Musculoskeletal and connective tissue disorders) | 15 (19) | 4 (4) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 13 (15) | 4 (4) | 4 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 16 (20) | 6 (8) | 6 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 26 (29) | 11 (15) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 9 (10) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 (48) | 14 (18) | 8 (17)
Dizziness (Nervous system disorders) | 37 (44) | 11 (12) | 6 (6)
Dysgeusia (Nervous system disorders) | 45 (48) | 18 (22) | 7 (8)
Headache (Nervous system disorders) | 31 (42) | 9 (10) | 5 (6)
Neuropathy peripheral (Nervous system disorders) | 9 (9) | 18 (20) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (8) | 11 (16) | 2 (2)
Taste disorder (Nervous system disorders) | 7 (7) | 7 (8) | 2 (2)
Insomnia (Psychiatric disorders) | 22 (23) | 14 (16) | 2 (2)
Haematuria (Renal and urinary disorders) | 15 (17) | 8 (9) | 4 (4)
Urinary retention (Renal and urinary disorders) | 5 (5) | 1 (1) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 17 (17) | 8 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45 (66) | 15 (21) | 6 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 26 (28) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 23 (24) | 10 (12) | 2 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 27 (39) | 0 (0) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (24) | 5 (9) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 19 (27) | 4 (4) | 5 (6)
Hot flush (Vascular disorders) | 17 (18) | 3 (5) | 3 (3)
Hypertension (Vascular disorders) | 18 (36) | 11 (16) | 5 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (2):
  • Study Protocol (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT02975934/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT02975934/SAP_001.pdf